CLINICAL TRIAL: NCT03162679
Title: Culture-sensitive Emotion Regulation Group Therapy for Traumatized Refugees: A Randomized Controlled Trial
Brief Title: Culture-sensitive Emotion Regulation Group Therapy for Traumatized Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: REFUGIO Munich (Unknown)
Responsible Party: Principal Investigator, Theresa Koch, Phd Student, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 022ERT
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Trauma
Keywords: trauma treatment; Refugees; Emotion regulation; Group therapy; randomized controlled; PTSD
MeSH Terms: conditions — Wounds and Injuries; Emotional Regulation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Regulation Group Therapy (Experimental): Participants assigned to this condition will receive treatment immediately after assignment.
  Interventions: Behavioral: Skills training of Affect-Regulation - A culture-sensitive approach: STARK
- Wait List Control (No Intervention): This condition is a wait-list control and receives no intervention during the study period, but is offered treatment after the final assessment directly after the treatment phase of the intervention group.

INTERVENTIONS:
Behavioral: Skills training of Affect-Regulation - A culture-sensitive approach: STARK — Emotion Regulation Group Therapy, 14 sessions, 1.5 hour sessions, group therapy, meeting weekly.
  Other Names: German title: Skills-Training der Affektregulation: Ein kultursensibler Ansatz: STARK
  Arms: Emotion Regulation Group Therapy

SUMMARY:
There is a lack of studies on treatment effect in traumatised refugees. Recent findings indicate that emotion regulation deficits play a key role in PTSD also among traumatized refugees and highlight the importance and potential directions for the development of an emotion regulation training for refugees. In this study, the investigators therefore want to examine the effectiveness of a new, transdiagnostic, cultural-sensitive group therapy, which systematically teaches specific emotion regulation strategies. Participants will be randomly assigned to either the emotion regulation training, delivered in group format or a wait list control condition. The study takes place in cooperation with REFUGIO Munich, which is a treatment centre specialised in the treatment of traumatised refugees. Clinicians will deliver the treatment to traumatized asylum seekers and refugees that report difficulties in emotion regulation. The investigators will examine if refugees and asylum seekers in the intervention group will show improvements in psychological symptoms, social functioning as well as in emotion regulation in comparison to a wait list control group which will receive the treatment after the intervention group has completed. The group therapy covers 14 sessions and has a cognitive-behavioural background. It focuses on conveying strategies to cope with intense feelings and the patients should gain a sense of self-efficacy and control over their trauma-relevant feelings and symptoms. Qualified interpreters will be used in the assessments as well as group therapies.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or asylum seeker from Afghanistan, speaking Dari
* reporting at least one traumatic event on a trauma list
* reporting difficulties in emotion regulation
* between the age of 15 and 21 years

Exclusion Criteria:

* Psychosis
* Serious suicidal ideations
* Currently receiving psychotherapy elsewhere
* Serious dissociation

Ages: 15 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Difficulties in Emotion Regulation | baseline, after 14 weeks (= post-treatment), 3-months-follow-up (3 months after the treatment)
  Scale: Emotion Regulation Scale (DERS)
Change in General Health | baseline, after 14 weeks (= post-treatment), 3-months-follow-up (3 months after the treatment)
  Scale General Health Questionnaire -28 (GHQ-28)

SECONDARY OUTCOMES:
Change in posttraumatic stress | baseline, after 14 weeks (= post-treatment), 3-months-follow-up (3 months after the treatment)
  Scale: PTSD Checklist for DSM-5 (PCL-5)
Change in Anger Reactions | baseline, after 14 weeks (= post-treatment), 3-months-follow-up (3 months after the treatment)
  Scale: Dimensions of Anger Reactions-5 (DAR-5)
Treatment Experience Scale - Patient (TESP) | after 14 weeks (= post-treatment)
Change in emotional competence (Third party assessment by caregiver) | baseline, after 14 weeks (= post-treatment), 3-months-follow-up (3 months after the treatment)
  Scale: Emotional Competence Questionnaire (German: Emotionale-Kompetenz-Fragebogen - Fremdbeurteilung (EKF))

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Liedl, PhD, Principal Investigator — REFUGIO München; Theresa Koch, M.Sc., Study Director — Ludwig-Maximilians-Universität München/ REFUGIO München; Thomas Ehring, Professor, Study Chair — Ludwig-Maximilians-Universität München
Locations (1):
- REFUGIO München, Munich, Germany